CLINICAL TRIAL: NCT03271138
Title: A Randomized Controlled Trial of Dietary Supplementation With Bifidobacterium Infantis NLS Super Strain Among Celiac Disease Patients on a Gluten-free Diet With Persistent Gastrointestinal Symptoms
Brief Title: Bifidobacterium Infantis NLS Super Strain for Celiac Disease Patients on a Gluten-free Diet With Persistent Gastrointestinal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Global Institute of Probiotics (Other)
Collaborators: Dr. C. Bonorino Udaondo Gastroenterology Hospital (Other Government); Research Institute, Universidad del Salvador (Unknown); Consejo de Investigaciones en Salud, Ministerio de Salud, Gobierno Autónomo de Buenos Aires (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: GlobalIP; 001 (Other Grant/Funding Number: Dr. C. Bonorino Udaondo Gastroenterology Hospital)
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Gluten-Free Diet; Bifidobacterium infantis NLS super strain; gastrointestinal symptoms; quality of life; microbiota; IgA TTG; IgA DGP
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bifidobacterium Infantis NLS Super Strain (Active Comparator): Participants in the probiotic period will take two capsules of Bifidobacterium infantis NLS super strain (Natren LIFE START®2) three times per day for three weeks. Each capsule contains 2 x 10^9 colony-forming units (CFU) of Bifidobacterium infantis NLS super strain, for a total daily dose of 12 X 10^9 CFU. The probiotic will be kept refrigerated during transportation and throughout the study period.
  Interventions: Dietary Supplement: Bifidobacterium infantis NLS super strain (Natren LIFE START®2)
- Placebo (Placebo Comparator): Participants in the placebo period will take two capsules of placebo three times per day for three weeks. The placebo capsules contain rice flour, hydroxypropyl and methylcellulose. The placebo will be kept refrigerated during transportation and throughout the study period.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium infantis NLS super strain (Natren LIFE START®2) — 2 capsules, 3 times per day, for daily total of 12x10^9 CFU Bifidobacterium infantis NLS super strain
  Arms: Bifidobacterium Infantis NLS Super Strain
Other: Placebo — 2 capsules, 3 times per day, containing rice flour, hydroxypropyl and methylcellulose
  Arms: Placebo

SUMMARY:
The primary purpose of this randomized, double-blinded, placebo-controlled, crossover clinical trial is to evaluate the efficacy of dietary supplementation with Bifidobacterium infantis NLS super strain among celiac disease patients on a gluten-free who have persistent gastrointestinal symptoms.

DETAILED DESCRIPTION:
Most patients with celiac disease demonstrate substantial clinical improvement during the first few weeks after the onset of the consumption of a gluten-free diet. However, between 30-50% of patients with celiac disease have persistent gastrointestinal symptoms despite consuming a gluten-free diet and presenting negative antibodies. It has recently been reported that celiac disease patients treated with a gluten-free diet that still have persistent symptoms possess different intestinal microbiota patterns than patients without persistent symptoms. Furthermore, a pilot study showed that dietary supplementation with probiotics (Bifidobacterium infantis NLS super strain - Natren LIFESTART®) in untreated celiac disease patients was associated with a significant improvement in symptoms as compared to placebo. Collectively, these findings contribute to the hypothesis that celiac disease patients on a gluten-free diet in whom gastrointestinal symptoms persist may benefit from the supplementation of Bifidobacterium infantis NLS super strain.

Participants in this double-blinded crossover trial will be randomized to receive either placebo or Bifidobacterium infantis NLS super strain for 3 weeks, followed by a 2 week washout period, and then followed by 3 weeks of the other of either placebo or probiotic supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women at least 18 years of age
* Precise diagnosis of celiac disease: serology (a-tTG IgA and/or DGP IgG and/or EmA) and histology (Marsh IIIa or greater) concordantly positive, confirmed at investigator's institution
* Consuming a gluten-free diet for at least 2 years
* Persistent gastrointestinal symptoms: global GSRS questionnaires ≥2 or ≥ 3 points for any of the 5 sub-dimensions
* Signature of informed consent

Exclusion Criteria:

* Patients not interested or unable to comply with questionnaires and collection of samples of blood, feces, and urine
* Complicated celiac disease (refractory, ulcerative jejunoileitis, lymphoma)
* Concomitant pathologies that are uncompensated or untreated (Type I or II diabetes mellitus, hyperthyroidism, hypothyroidism, diarrhea due to bile salts, pancreatic insufficiency, bacterial overgrowth)
* Consumption within the 2 weeks prior to study enrollment of medication that interferes with bowel functioning (antibiotics, NSAIDs, laxatives, metformin, opiates, anticholinergics [atropine, antidepressants, neuroleptics, antipsychotics, antiparkinsonians], anticonvulsants, antihistamines, antihypertensives [calcium antagonists, clonidine, diuretics, metal ions (aluminum), antacids, sucralfate, barium sulfate, bismuth, calcium, iron, heavy metals (arsenic, lead, mercury)], resins (cholestyramine), or any other medication deemed relevant by the investigator).
* Women that are pregnant or may become pregnant during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-07-21 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Changes in Gastrointestinal Symptom Rating Scale (GSRS) | Baseline, End of Period I (3 weeks), End of Period II (8 weeks)

SECONDARY OUTCOMES:
Changes in Celiac Symptoms Index (CSI) | Baseline, End of Period I (3 weeks), End of Period II (8 weeks)
Changes in Quality of Life: SF-36 | Baseline, End of Period I (3 weeks), End of Period II (8 weeks)
Changes in gut microbiota | Baseline, End of Period I (3 weeks), End of Period II (8 weeks)
  16S rRNA Illumina based sequencing
Changes in Gluten Immunogenic Peptides (GIP) | Baseline, End of Period I (3 weeks), End of Period II (8 weeks)
Changes in serology (IgA tTG & IgA DGP) | Baseline, End of Period I (3 weeks), End of Period II (8 weeks)
Changes in anthropometric measurements (BMI) | Baseline, End of Period I (3 weeks), End of Period II (8 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Edgardo Smecuol, MD, Principal Investigator — Dr. C. Bonorino Udaondo Gastroenterology Hospital; Julio C Bai, MD, Study Director — Dr. C. Bonorino Udaondo Gastroenterology Hospital
Locations (1):
- Small Bowel Section, Department of Medicine, Dr. C. Bonorino Udaondo Gastroenterology Hospital, Buenos Aires, Argentina

REFERENCES:
- [Derived] Smecuol E, Constante M, Temprano MP, Costa AF, Moreno ML, Pinto-Sanchez MI, Vazquez H, Stefanolo JP, Gonzalez AF, D'Adamo CR, Niveloni SI, Maurino E, Verdu EF, Bai JC. Effect of Bifidobacterium infantis NLS super strain in symptomatic coeliac disease patients on long-term gluten-free diet - an exploratory study. Benef Microbes. 2020 Oct 12;11(6):527-534. doi: 10.3920/BM2020.0016. Epub 2020 Oct 9. PMID 33032471